CLINICAL TRIAL: NCT06914271
Title: Effects of Kendall Exercises Versus Kabat Exercises in Patients With Chronic Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/819
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kendall Exercise (Experimental)
  Interventions: Combination Product: Kendall Exercise
- Kabat Exercises (Active Comparator)
  Interventions: Combination Product: Kabat Exercises

INTERVENTIONS:
Combination Product: Kendall Exercise — The Kendall Exercises focus on correcting posture, strengthening the core, and re-educating muscles to improve spinal alignment and reduce pain .These exercises primarily target specific muscles and joint actions to help patients regain their range of motion.
  Arms: Kendall Exercise
Combination Product: Kabat Exercises — The principle of the Kabat exercises is based on a series of neuromuscular facilitation techniques that emphasize dynamic movement patterns, flexibility, and coordination to enhance functional mobility and alleviate pain.
  Arms: Kabat Exercises

SUMMARY:
Low back pain (LBP) is pain, muscle tension, or stiffness under the costal border and above the inferior gluteal folds, with or without leg pain.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Adults Aged Between 30-65
* Low Back pain should be Persistent for more than 12 weeks
* Visual Analogue scale or VAS of 3 or higher
* Idiopathic pain
* Ability to engage in physical activity and participate in the intervention program
* Willingness and ability to provide informed consent to participate in the study

Exclusion Criteria:

* Low back pain due to other causes

  1. Fibromyalgia
  2. Previous spine surgery
  3. Spondylolisthesis
  4. Spondylolysis
  5. Rheumatoid arthritis or Ankylosing spondylitis
  6. Spinal inflammation or tumor
  7. Spinal or pelvis fracture
  8. Osteoporosis
  9. Respiratory or heart diseases
  10. Stroke
  11. Pregnancy
* Persistent use of pain medication
* Patients who had undergone any other treatments, such as acupuncture or physical therapy, in the last 3 months
* Anticipated inability to comply with study protocols or attend scheduled."

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12 Months
  The Visual Analogue Scale (VAS) is a way of measuring pain intensity. It is often utilized in investigations concerning pain management. Visual analog scales (VAS) are psychometric measuring tools created to record the characteristics of disease-related symptom severity in individual patients and utilize this to achieve a quick (statistically observable and reproducible) classification of symptom severity and disease control. Scores are taken by placing a handwritten mark along a 10-cm line that depicts a pain spectrum between ""no pain"" and ""worst pain.""
Oswestry Disability Index (ODI) | 12 Months
  The Oswestry Disability Index (ODI) is a widely used instrument for determining the degree of impairment and how low back pain affects a person's ability to do daily chores. Each of its 10 sections focuses on a different aspect of everyday life, such as pain severity, personal cleanliness, walking, lifting, sitting, standing, sleeping, and social life. A person's scores for each component are added based on the severity of their condition to determine their total disability percentage, which can range from 0% (no impairment) to 100% (severe disability). It is widely used in clinical settings to track changes over time and assess the effectiveness of treatments for low back pain (27).
  The Oswestry Disability Index (ODI) exhibits great validity (correlation with VAS: r= 0.67; Roland Morris: r=0.76) and high reliability (Cronbach's α > 0.70, ICC > 0.90)
Goniometer | 12 Months
  A Goniometer is simple yet effective tool used to measure the range of motion of a joint.
  0% to 20%: minimal disability:
  21%-40%: moderate disability: 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation.
  61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required.
  81%-100%: These patients are either bed-bound or exaggerating their symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Younas hospital daska, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No